CLINICAL TRIAL: NCT04954443
Title: Urinary Retention After Removing Urinary Catheter at 24 Hour Comparison With 48 Hour in Patients With Vaginal Surgery of Pelvic Organ Prolapse, Randomized Controlled Trial
Brief Title: Urinary Retention After Removing Urinary Catheter at 24 Hour Versus 48 Hour in Patients With Vaginal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 084/2564
Record Dates: First submitted 2021-05-12; First posted 2021-07-08 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Urinary Retention; Pelvic Organ Prolapse
Keywords: Urinary Retention; Pelvic Organ Prolapse; Vaginal surgery; Urinary catheter
MeSH Terms: conditions — Urinary Retention; Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Single blind (Care provider, investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Removing urinary catheter at 24 hours after surgery (Experimental): The participants will removing urinary catheters at 24 hour after vaginal surgery of pelvic organ prolapse.
  Interventions: Procedure: Removing urinary catheter
- Removing urinary catheter at 48 hours after surgery (Placebo Comparator): The participants will removing urinary catheters at 48 hour after vaginal surgery of pelvic organ prolapse.
  Interventions: Procedure: Removing urinary catheter

INTERVENTIONS:
Procedure: Removing urinary catheter — Removing urinary catheter after vaginal surgery of pelvic organ prolapse

SUMMARY:
Comparison incident of urinary retention in patients with vaginal surgery of pelvic organ prolapse, who removed urinary catheter at 24 hours versus 48 hours after surgery

DETAILED DESCRIPTION:
Vaginal surgery of pelvic organ prolapse needs to insert urinary catheter for monitoring post-operative complication, hemodynamic status, and prevention post-operative urinary retention. Urinary retention occur 2.4 - 43% after pelvic organ prolapse surgery, whereas retaining urinary catheter is common cause of urinary tract infection, often hospital-acquired infection. At Rajavithi hospital always remove urinary catheter at 48 hour after surgery. Accordingly, appropriated time for removing urinary catheter in patients with vaginal surgery of pelvic organ prolapse is unclear. This study aims to reduce timing for removing urinary catheter after vaginal surgery, not increase urinary retention and re-catheterization and reduce urinary tract infection and day of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Woman with pelvic organ prolapse, who undergoing vaginal surgery and agrees to participate in this study
* Able to understand and communicate Thai language

Exclusion Criteria:

* Woman with diabetes mellitus with HbA1C > 10.9%
* Woman with stroke
* Woman with urinary tract infection before surgery
* Woman with urinary retention before surgery
* Woman, who experienced surgery for urinary incontinence
* Woman, with operative complication including of hemorrhagic shock (Blood pressure < 90/60 mmHg, Heart rate > 120 beats per minute, Intra-operative blood loss > or = 750 ml), urinary tract injury, bowel injury

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Urinary retention | Through study completion, an average of 1 year
  Incident of urinary retention (Post-void residual urine at least 150 ml) after removing urinary catheter at 24 hour comparison with 48 hour after vaginal surgery of pelvic organ prolapse

SECONDARY OUTCOMES:
Re-catheterization after removing urinary catheter | Through study completion, an average of 1 year
  Incident of re-catheterization after removing urinary catheter at 24 hour comparison with 48 hour after vaginal surgery of pelvic organ prolapse
Urinary tract infection | Through study completion, an average of 1 year
  Incident of urinary tract infection (positive urine culture) after removing urinary catheter at 24 hour comparison with 48 hour after vaginal surgery of pelvic organ prolapse

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand